CLINICAL TRIAL: NCT05600257
Title: The Effect of Digital Breast Tomosynthesis in Breast Cancer Long-term Survival: a Single Institution Study
Status: Completed | Type: Observational
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Chen-Pin Chou, Radiologist, Kaohsiung Veterans General Hospital.
Other Study IDs: KSVGH22-CT11-01
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening cohort: Women received mammography screening
  Interventions: Device: DBT; Device: DM
- Diagnostic cohort: Women received clinical breast examination
  Interventions: Device: DBT; Device: DM

INTERVENTIONS:
Device: DBT — Image with digital breast tomosynthesis
  Other Names: Digital Breast Tomosynthesis
Device: DM — Image with digital mammography
  Other Names: Digital Mammography

SUMMARY:
To investigate whether digital breast tomosynthesis (DBT) benefits survival improvement.

DETAILED DESCRIPTION:
To suggest DBT for specific populations, compare the overall survival rate of women with digital mammography (DM) to the DBT screening for women with particular characteristics.

ELIGIBILITY:
Inclusion Criteria:

* individuals were diagnosed with breast cancer according to the International Disease Classification Criteria

Exclusion Criteria:

* no surgery or incomplete surgical pathology stage
* complete remission after neoadjuvant chemotherapy
* non-breast cancer death
* bilateral breast cancer
* male breast cancer
* no pre-surgery mammography image

Ages: 23 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals were diagnosed with breast cancer according to the International Disease Classification Criteria from September 2011 to December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 1517 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Overall survival rate | Up to 111 months
  Compare the overall survival rate according to breast density type, cancer stage, mammography test type, and imaging modality.

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Pin Chou, MD, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on reasonable request from the corresponding author. Some data are not publicly available due to their containing information that could compromise the privacy of research participants.